CLINICAL TRIAL: NCT05294510
Title: STewardship for Acute Respiratory Illness (STAR): a Stepped Wedge, Cluster Randomized Trial of Point-of-care Biomarker Testing by Village Health Workers
Brief Title: Improving Antibiotic Stewardship for Children With Respiratory Illness Presenting to Village Health Workers in Uganda
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-2803; 15206 (Other Grant/Funding Number: Thrasher Research Fund)
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Infections in Children
Keywords: Community health workers; C-reactive protein

STUDY DESIGN:
Intervention Model Description: Stepped wedge, cluster randomized trial with 5 clusters or treatment sequences of 3 villages each. Villages are first stratified by altitude, proximity to the local health center, and size (based on approximate number of children seen by the village health workers per year) into one of three strata: (1) low altitude, proximal, large, (2) low altitude, mid-distance, medium, (3) high altitude, distal, small. One village is then randomly selected from each strata for each of the 5 clusters. All clusters start in the control condition and one cluster crosses over from control to intervention each month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Children who present to a village health worker during a control period are evaluated and managed using the current standard of care per Uganda National Guidelines for Integrated Community Case Management (ICCM). Each village will experience both Control and Intervention conditions as the study employs a stepped wedge design.
- Intervention (Experimental): Children who present to a village health worker during an intervention period are evaluated and managed using a modified ICCM algorithm that includes point-of-care C-reactive protein testing. Each village will experience both Control and Intervention conditions as the study employs a stepped wedge design.
  Interventions: Other: STAR Sick Child Job Aid

INTERVENTIONS:
Other: STAR Sick Child Job Aid — The STAR Sick Child Job Aid is a modified ICCM protocol that includes the addition of a point-of-care C-reactive protein (CRP) test to inform antibiotic treatment decisions for children presenting with febrile acute respiratory illness who do not have any danger signs. If CRP ≥ 40 mg/L, the village health worker (VHW) will dispense amoxicillin per local guidelines. If CRP < 40 mg/L, the VHW will advise symptomatic care alone including acetaminophen for fever and additional fluids to maintain hydration.
  Arms: Intervention

SUMMARY:
This is a stepped wedge, cluster randomized study of a clinical algorithm that includes point-of-care C-reactive protein testing to inform antibiotic treatment decisions by village health workers for children presenting with acute respiratory illness in the Bugoye sub-county of the Kasese District in southwestern Uganda.

The purpose of this study is to assess the impact of the algorithm on antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 months-5 years
* Evaluated by a study VHW in one of the participating villages in Bugoye sub-county for acute respiratory illness defined as the following: fever (documented (temperature > 38°C) or subjective fever in the last seven days) AND fast breathing (respiratory rate > 30) OR cough

Exclusion Criteria:

* Age > 5 years or < 2 months at time of presentation
* Guardian not present to provide consent

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1280 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescriptions at baseline visit | Baseline visit
  Proportion of children prescribed antibiotics by the village health worker at the baseline visit in the control as compared to the intervention condition.

SECONDARY OUTCOMES:
Clinical Failure (Composite Outcome) | Between baseline visit and Day 7 follow-up assessment
  Proportion of children with one or more of the following outcomes in the control as compared to the intervention condition: persistence of fever at Day 7, development of danger signs as defined by local Integrated Community Care Management guidelines at any time during the seven-day follow-up period, need for hospitalization at any time during follow-up period, or death at any time during follow-up period.
Unexpected visits | Between baseline visit and Day 7 follow-up assessment
  Proportion of children brought to the village health worker during the seven-day follow-up period for persistent or worsening symptoms by their caregiver in the control as compared to the intervention condition.
Perceived improvement per caregiver | Day 7
  Proportion of caregivers who perceive that their child has clinically improved at the Day 7 follow-up assessment in the control as compared to the intervention condition.
Persistent fever | Day 7
  Proportion of children who have persistence of subjective or documented fever at the Day 7 follow-up assessment in the control as compared to the intervention condition.
Development of danger signs | Between Day 1 and Day 7
  Proportion of children who develop danger signs (as defined by local Integrated Community Care Management guidelines) during the seven-day follow-up period in the control as compared to intervention conditions.
Hospitalization | Between Day 1 and Day 7
  Proportion of children who require inpatient admission to a health facility during the seven-day follow-up period in the control as compared to intervention periods.
Death | Between Day 1 and Day 7
  Proportion of children who die during the seven-day follow-up period in the control as compared to intervention periods.
Antibiotic prescriptions during study follow-up | Between baseline visit and Day 7 follow-up assessment
  Proportion of children prescribed antibiotics by any provider either at the baseline visit or during the seven-day follow-up period in the control as compared to the intervention condition.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Ciccone, MD, MHS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bugoye Health Center III, Bugoye, Kasese District, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that underlie the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 9 months to 36 months after publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC

REFERENCES:
- [Derived] Ciccone EJ, Hu D, Preisser JS, Cassidy CA, Kabugho L, Emmanuel B, Kibaba G, Mwebembezi F, Juliano JJ, Mulogo EM, Boyce RM. Point-of-care C-reactive protein measurement by community health workers safely reduces antimicrobial use among children with respiratory illness in rural Uganda: A stepped wedge cluster randomized trial. PLoS Med. 2024 Aug 19;21(8):e1004416. doi: 10.1371/journal.pmed.1004416. eCollection 2024 Aug. PMID 39159269